CLINICAL TRIAL: NCT03531359
Title: Tablet-based Interactive Distraction for the Management of Preoperative Anxiety in Children: A Randomized Controlled Trial
Brief Title: Tablet-based Interactive Distraction Preoperative Anxiety in Children: A Randomized Controlled Trial
Acronym: TABLET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Hospital Carlos Van Buren (Other)
Responsible Party: Principal Investigator, Nathalie Lopez, Principal Investigator, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV-1-2018
Record Dates: First submitted 2018-04-30; First posted 2018-05-21 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Children Under General Anaesthesia
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Tablet Group: They'll receive a tablet with content adapted to every group. It will be divided into 4 groups (2-4 years, 4-6 years, 6-8 years and 9-10 years). The first one will receive cartoons, the second will also have games; for the other two groups will be assigned appropriate video games depending on the age.
  Midazolam group: They'll receive 0,5mg/kg oral or it's equivalent in rectal administration 30 minutes to one hour prior to transfer to the theater. This patients will not be able to have contact with audiovisual devices.
Who Masked: Outcomes Assessor
Masking Description: Anxiety will be determined by using a video recording of the child, which will be assessed by psychiatric
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIBD Tablet-based video distraction (Experimental): Children will receive of tablet-based interctive games in preoperatory room
  Interventions: Device: TIBD
- Midazolam (Active Comparator): Children will be premedicated with usual treatmente (midazolam)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Device: TIBD — Table-based Interactive Distraction using video-games will be used to prove efficacy in preventing preoperative anxiety.
  Arms: TIBD Tablet-based video distraction
Drug: Midazolam — Administration of midazolam oral or rectal 30 minutes to one hour prior to transfer to the theater.
  Arms: Midazolam

SUMMARY:
Children develop anxiety during the induction of anaesthesia and video-games might reduce or alleviate it. The investigators intend to conduct a clinical trial to study the effect of tablet-based interctive games on alleviating preoperative anxiety.

DETAILED DESCRIPTION:
It is estimated that 50% of children may suffer preoperative anxiety. They have a higher risk of generating postanesthetic delirium and behavioral changes in the postoperative period up to 67% of cases.

For the management of preoperative anxiety there are pharmacological and non-pharmacological treatments. Within the first group there's the use of benzodiazepines of short half life like midazolam, however, the use of this medication is not exempt of risks such as paradox reactions, respiratory depression, among others. This is why the non pharmacological mesures have taken force and every day there is more evidence regarding its effectiveness.

There are no reports in Chile or latin america regarding the use of this tools, this is why the investigators designed this study to prove the effectiveness of audiovisual distraction measures in reducing preparatory anxiety compared to premeditation with midazolam.

ELIGIBILITY:
Inclusion Criteria:

Children aged 2-10 years, under major surgery ambulatory program at Hospital Carlos Van Buren, with no contraindication for the use of midazolam.

Exclusion Criteria:

Patients with cognitive impairment or sensory deficit Patients with previous history of major surgery will also be excluded Patients with myastenia "Hard airway" History of paroxystic reaction to benzodiazepines Attentional deficit hyperactivity disorder Sleep aphnea Full stomach Adenotonsillar hypertrophy Respiratory acute infections

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Short version of the modified Yale Preoperative Anxiety Scale(mYPAS-SF) | 6 hours
  Difference between the measurement of the mYPAS-SF applied in the preoperative time and prior to induction.
  The scale has 18 items in 4 categories. Maximum score is 100 points. The higher the score, the greater the anxiety.

SECONDARY OUTCOMES:
Cooperation with the induction | 30 minuts
  Scale with 10 items, 1 point for each one. 0 points shows an induction with perfect cooperation.
  This scale will be applied at the moment of the induction by the anesthesiologist
Changes in postoperative behavior | 10 days
  The Post Behavioral Behavior Change Questionnaire (PHBQ) will be applied at the postoperative surgical control (7-10 days after the intervention). This survey will be applied by people trained by the hospital's pediatric psychiatry team The higher the score, the more behavioral changes in the postoperative period
Emergence delirium | 1 hour
  In the post-anesthesia recovery unit, the Emergency Delirium Scale for Pediatric Anesthesia (PAED) will be applied every 15 minutes during the first 30 minutes of their stay in the unit. Score goes from 0 to 20. Scores greater than 10 is considered as delirium.
Parents Satisfaction | 10 minuts
  A gradual scale will be applied to the parents of the patient upon discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie López, MD, Study Director — Universidad de Valparaíso Chile; Anamaria Correa, MD, Principal Investigator — Universidad de Valparaíso Chile
Locations (1):
- Hospital Carlos Van Buren, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided